CLINICAL TRIAL: NCT05545605
Title: Efficacy and Safety of Sodium Oligomannate in the Prevention of Post-stroke Cognitive Impairment in Patients With Ischemic Stroke:a Randomized, Double-blind, Exploratory Controlled Study
Brief Title: Efficacy and Safety of Sodium Oligomannate in the Prevention of PSCI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NFEC-2022-276
Record Dates: First submitted 2022-09-15; First posted 2022-09-19 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Ischemic Stroke
Keywords: Post-stroke cognitive impairment; gut microbiota; Sodium oligomannate
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Statistical researchers from the partner Shanghai Green Valley Pharmaceutical Co., LTD., used statistical software packages to generate two sets of 58 random drug numbers, which were determined in the form of files after the codes were formed.Masking the participant and investigator.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Subjects randomized to the trial group will receive sodium oligomannate 450mg twice daily for 24 weeks.
  Interventions: Drug: Sodium oligomannate
- Control group (Placebo Comparator): Subjects randomized to the control group will receive a 450mg placebo capsule twice daily for 24 weeks that has exactly the same appearance and smell as the Intervention group.
  Interventions: Drug: Placebo capsule

INTERVENTIONS:
Drug: Sodium oligomannate — Patients with acute ischemic stroke were recruited, and after signing informed consent, those who met the inclusion/exclusion criteria were randomly assigned in a 1:1 ratio to receive treatment in the trial group (receiving sodium oligomannate)
  Arms: Intervention group
Drug: Placebo capsule — the control group (receiving placebo capsule) for 24 weeks.
  Arms: Control group

SUMMARY:
Post-stroke cognitive impairment (PSCI) is a common complication of stroke, and seriously affect the quality of survival and the survival time in patients with stroke, PSCI is still lack of effective prevention and treatment measures, the study found that gut microbiota are closely associated with stroke and cognitive diseases, sodium oligomannate can improve cognitive function of mild-to-moderate alzheimer's disease (AD) , The Expert Consensus 2021 on the Management of Post-stroke cognitive impairment states that the role of sodium oligomannate in PSCI needs to be investigated in large sample clinical trials. This study intends to explore the efficacy and safety of sodium oligomannate in the prevention of PSCI in patients with acute ischemic stroke and cognitive impairment, so as to provide a potential intervention for the prevention of PSCI.

DETAILED DESCRIPTION:
This clinical study was a randomized (1:1), double-blind, single-center, parallel controlled clinical study. The study period was 6 months to evaluate the efficacy and safety of sodium oligomannate in the prevention of PSCI in patients with ischemic stroke. Patients with acute ischemic stroke were recruited. After signing informed consent, patients who met the inclusion/exclusion criteria were randomly assigned in a 1:1 ratio to receive treatment in the trial group (receiving sodium oligomannate) or the control group (receiving placebo capsule). A total of 116 patients were enrolled.And safety assessment and survival follow-up were performed at 4 weeks, 12 weeks and 24 weeks, and efficacy assessment was performed at 12 weeks and 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* 1.The first occurrence of ischemic stroke, which met the diagnostic criteria of the Chinese Guidelines for the Diagnosis and Treatment of Acute Ischemic Stroke 2018, was confirmed by CT or MR; 2. The onset of illness was less than 7 days after admission, aged 18-80 years; 3. Clear consciousness, able to cooperate with cognitive and other tests, NIHSS score ≤15; 4. Before onset, the patient's cognitive level was normal, daily life and social activities were normal; 5. Stay in the current place of residence for more than 3 years; 6. With cognitive assessment, MoCA < 22 (years of education < 12, +1) after correction, and signed the informed consent.

Exclusion Criteria:

* 1.Unable to cooperate with neuropsychological examination due to various reasons (such as consciousness disorders, vision disorders, hearing disorders, etc.); 2. Combined with other diseases (such as intracranial mass, demyelinating disease, intracranial infection, neurodegenerative disease, epilepsy, severe heart, liver, kidney, blood system or other system diseases, etc.); 3. Used antibiotics 3 months before onset; 4. A history of alcohol abuse, drug use, or serious mental illness (including major depression (HAMD > 10)) before onset of illness, 5. No stool was collected within 7 days of onset.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of PSCI | 6 months
  Proportion of patients in both groups with a corrected MoCA score of < 22 at 24 weeks of medication

SECONDARY OUTCOMES:
Incidence of adverse events | 6 months
  The proportion of patients who had any adverse effect during the study period
The difference of MoCA value from cardinality | 6 months
  The difference between the MoCA value at 24 weeks of medication and the MoCA value at enrollment
Differences in ADAS-cog values from cardinality | 6 months
  The difference between the ADAS-cog value at 24 weeks of medication and the ADAS-cog value at enrollment.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Nanfang Hospital, Southern Medical University, Guangzhou, Baiyun
  - Nanfang Hospital,Southern Medical University, Guangzhou, Guangdong

IPD SHARING:
Plan to Share IPD: Undecided